CLINICAL TRIAL: NCT00700609
Title: Family-Based Treatment of Depressed Adolescents: An Empirical Study With Norwegian Adolescents in Specialty Mental Health Care
Brief Title: Family Based Treatment of Depressed Adolescents
Acronym: BudFam
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The PI moved to another city and position
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18651
Record Dates: First submitted 2008-06-13; First posted 2008-06-18 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Depressive Disorder; Mood Disorder; Major Depression
Keywords: Depression; Family Therapy; Adolescents
MeSH Terms: conditions — Depressive Disorder; Mood Disorders; Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Attachment Based Family Therapy (ABFT)
  ABFT developed by Dr. Guy Diamond and colleagues is a brief, 12 week, manualized family-based intervention.
  Interventions: Behavioral: Attachment Based Family therapy (ABFT)
- 2 (Active Comparator): Treatment as usual (TAU)
  No attempt is made to standardize TAU. Regular clinical staff will provide mental health services.
  Interventions: Behavioral: Attachment Based Family therapy (ABFT)

INTERVENTIONS:
Behavioral: Attachment Based Family therapy (ABFT) — Attachment-Based Family Therapy (ABFT) is a brief manualized therapy designed exclusively for depressed adolescents and aims at reducing adolescent depression by improving family communication and trust.
  Other Names: ABFT; TAU

SUMMARY:
The purpose of this project is to assess the effectiveness of a family-based therapy (Attachment based family therapy-ABFT) for Norwegian adolescents (13-17 years) referred to specialist mental heath clinics.

DETAILED DESCRIPTION:
Depression is a major public health concern among adolescents. Research suggests that it not only is prevalent among adolescents (as many as 20% of adolescents have a depressive episode by the age of 18), but its effects last well into adulthood. Although available studies of psychosocial and pharmacological interventions show promise, there are concerns regarding their effectiveness and possible side effects like increase in suicidal ideation. Family conflict is not only an effect of depression, but also a risk factor for depression. High conflict and dysfunction, have consistently been shown to increase risk for depression. As such, family treatments that target risk and protective factors (e.g., quality of parent-child interaction, parental monitoring) for depression seem promising to reduce depression. The current study is a randomized clinical trail aimed at assessing the effectiveness of a 12-week family based intervention for depressed adolescents (Attachment based family therapy- ABFT). Adolescents referred to specialist mental health hospital in south-west Norway (Stavanger University Hospital) will be randomized to either ABFT or treatment as usual (TAU). Therapists administering both the experimental and control group intervention are regular staff clinicians. Outcome assessments would be carried out at baseline, 6, 12 and 26 weeks by raters blind to the condition of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* 13-17 years
* Referred to specialist mental health hospital
* HAM-D score of >14
* Meets diagnostic criteria for major depressive disorder or depression NOS
* Have a parent or guardian willing to participate

Exclusion Criteria:

* Suicidal and require in-patient care
* Low intellectual abilities
* Current psychosis
* primary caregiver unwilling to participate

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2008-06; Primary Completion 2009-03 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating scale (HAM-D, 17 items) | Baseline, 6, 12 and 26 weeks

SECONDARY OUTCOMES:
Beck depression Inventory (BDI-II) | Bi-weekly for 12 weeks
Kiddie- SADS (diagnostic interview) | Baseline and 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pravin Israel, Ph.D, Principal Investigator — Helse Stavanger HF
Locations (1):
- Department of Child and Adolescent Psychiatry, Stavanger University Hospital, Stavanger, Rogaland, Norway